CLINICAL TRIAL: NCT06994039
Title: The Comparative Study on Left Lateral Position and Supine Position in Endoscopic Ultrasound Guided Portal Pressure Gradient Measurement
Brief Title: Left Lateral Position and Supine Position in EUS-PPG Measurement
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0729
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05

CONDITIONS: Portal Pressure Gradient (PPG) Measurement Guided by Endoscopic Ultrasound (EUS); Left Lateral Decubitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EUS-suPPG: EUS-PPG measured in supine position
  Interventions: Procedure: EUS-lePPG

INTERVENTIONS:
Procedure: EUS-lePPG — EUS-PPG measured in left lateral decubitus position

SUMMARY:
The consistency of EUS-PPG measurements between left lateral decubitus and supine positions is unclear. In this prospective comparative study, we are aimed to evaluate the correlation between EUS-PPG measured in supine position (EUS-suPPG), and EUS-PPG measured in left lateral decubitus position (EUS-lePPG).

DETAILED DESCRIPTION:
The hepatic venous pressure gradient (HVPG) remains the gold standard for assessing portal hypertension, yet its clinical application faces several limitations. First, HVPG has restricted diagnostic scope, being unable to accurately evaluate prehepatic or presinusoidal portal hypertension. Second, the measurement process exposes both patients and physicians to radiation and involves complex techniques that preclude routine implementation in many hospitals. Finally, as HVPG indirectly estimates portal pressure through wedged hepatic venous pressure, its accuracy may be compromised by multiple factors including intrahepatic venous shunting, catheter insertion depth, excessive sedation or patient agitation during the procedure, and incomplete balloon occlusion of hepatic venous flow.

Endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) measurement effectively addresses these limitations of HVPG. Current clinical studies on EUS-PPG have predominantly been conducted in the supine position. However, this position significantly increases the technical difficulty of endoscopic ultrasonography and complicates the simultaneous performance of endoscopic selective varices devascularization (EUS-ESVD) under single anesthesia. The consistency of EUS-PPG measurements between left lateral decubitus and supine positions requires further investigation.

This prospective comparative study enrolls hospitalized patients with liver cirrhosis. EUS-guided puncture of both the portal vein and hepatic vein were performed using a 25G needle. Pressure transducers measure the portal venous pressure (PVP) and hepatic venous pressure (HVP), with their differential defined as EUS-PPG. Measurements obtained in supine position are designated EUS-suPPG, while those in left lateral decubitus position are termed EUS-lePPG. Statistical analysis will evaluate the correlation between EUS-suPPG and EUS-lePPG values, with postoperative monitoring for complications including infection and hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients with liver cirrhosis, and are willing to sign the informed consent.

Exclusion Criteria:

1. Unwilling to sign the informed consent
2. Severe coagulopathy (INR>1.6)
3. Severe thrombocytopenia (platelets <20,000/μL)
4. Bacteremia
5. Age<18, or≥81
6. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
EUS-lePPG | From the begining of zero calibration for pressure transducer to the end of the endoscopic procedure, until up to 1 day.
  EUS-PPG measured in left lateral decubitus position

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No